CLINICAL TRIAL: NCT04446741
Title: Developing a Molecular Diagnostic Platform for Personalized Medicine for Acute Myeloid Leukemia
Brief Title: Molecular Diagnostic Platform for AML
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PCR-LMA
Record Dates: First submitted 2020-06-17; First posted 2020-06-25 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: AML; Adult; Molecular
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow and peripheral blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Myeloid Leukemia (AML): Newly diagnosed or relapsed/resistant AML

SUMMARY:
This will be a translational study without any therapeutic intervention, for the purpose of analyzing the diagnostic and molecular results / characterization of adult patients with AML, regardless of the treatment they receive. Newly diagnosed or relapsed/resistant AML patients will be included.

DETAILED DESCRIPTION:
This will be a multicenter, translational study without any therapeutic intervention. It will be conducted at 7 central laboratories (Hospital Universitari i Politècnic La Fe, Hospital Universitario de Salamanca, Hospital 12 de Octubre, Hospital Universitario Virgen del Rocío, Hospital Dr. Negrín de Las Palmas de Gran Canaria, Hospital Reina Sofía de Córdoba and Clínica Universidad de Navarra) belonging to the Spanish PETHEMA Group. The laboratories will receive and process bone marrow and peripheral blood samples of patients with AML at the time of the initial diagnosis or at relapse or resistance (first or subsequent relapse/resistance). The demographic data and clinical characteristics of the patients and of the AML, morphological and molecular response will be collected in case report forms (CRFs). Since the aim of this study is the molecular diagnosis of AML, all patients with AML will be included, regardless of the treatment (or no treatment at all) they receive.

The physicians will receive the report about the molecular diagnosis for FLT3, NPM1, CBF and PML/RARa quickly (<48-96 hours), in order to provide them with knowledge of the mutational status, that may cause changes to be made during the initial management of the disease.

The aim of this project is to set up this rapid screening and diagnostic platform for AML by having specimens sent to 7 centralized reference laboratories across the country, where the molecular characteristics of leukemic cells will be analyzed by qRT-PCR and NGS technologies with high quality standards. This platform will provide homogeneous criteria for assessing the biological characteristics of the different entities that make up the disease.

It is expected that samples of marrow and/or blood of 700 patients with AML will be analyzed per year.

ELIGIBILITY:
Inclusion Criteria:

* Have voluntarily given informed consent for the sending and processing of biological specimens, as well as for the analysis and reporting of the results on the mutation status of their AML.
* Age greater than or equal to 18 years.
* Morphological diagnosis of AML or acute leukemia of ambiguous lineage according to WHO criteria at diagnosis, relapse or resistance.

Exclusion Criteria:

* Inability of the patient or his/her legal representative to understand and voluntarily sign the informed consent form

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years with a diagnosis of AML (new, relapse or refractory).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of FLT3, NPM1 and CEBPa mutations | Baseline
  Frequency of each of the standard screening panel molecular alterations studied in the AML patients (FLT3, NPM1 and CEBPa), both in newly diagnosed and relapsed/resistant disease.

SECONDARY OUTCOMES:
Frequency of mutations detected by Next Generation Sequency (NGS) | Baseline
  Frequency of mutations detected by NGS PCR (23 genes: FLT3, NPM1, DNMT3A, IDH2, IDH1, TET2, RUNX1, TP53, NRAS, WT1, PTPN11, KIT, U2AF1, KRAS, SMC1A, SMC3, PHF6, STAG2, RAD21, FAM5C, EZH2 and HNRNPK; if new genes are described,the panel can be extended) in every sample (diagnosis, relapse)
Frequency of mutations detected by conventional PCR (FLT3, NPM1 and CEBPa) in every sample (diagnosis, relapse) | Baseline
  Frequency of each of the standard screening panel molecular alterations studied by the conventional PCR in the AML patients (FLT3, NPM1 and CEBPa), both in newly diagnosed and relapsed/resistant disease.

CONTACTS AND LOCATIONS:
Overall Officials: Pau Montesinos, Principal Investigator — Hospital Universitario La Fe
Locations (7):
- Spain (7):
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital Doce de Octubre, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario La Fe, Valencia

REFERENCES:
- [Background] Dohner H, Estey EH, Amadori S, Appelbaum FR, Buchner T, Burnett AK, Dombret H, Fenaux P, Grimwade D, Larson RA, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz MA, Sierra J, Tallman MS, Lowenberg B, Bloomfield CD; European LeukemiaNet. Diagnosis and management of acute myeloid leukemia in adults: recommendations from an international expert panel, on behalf of the European LeukemiaNet. Blood. 2010 Jan 21;115(3):453-74. doi: 10.1182/blood-2009-07-235358. Epub 2009 Oct 30. PMID 19880497
- [Background] Ley TJ, Mardis ER, Ding L, Fulton B, McLellan MD, Chen K, Dooling D, Dunford-Shore BH, McGrath S, Hickenbotham M, Cook L, Abbott R, Larson DE, Koboldt DC, Pohl C, Smith S, Hawkins A, Abbott S, Locke D, Hillier LW, Miner T, Fulton L, Magrini V, Wylie T, Glasscock J, Conyers J, Sander N, Shi X, Osborne JR, Minx P, Gordon D, Chinwalla A, Zhao Y, Ries RE, Payton JE, Westervelt P, Tomasson MH, Watson M, Baty J, Ivanovich J, Heath S, Shannon WD, Nagarajan R, Walter MJ, Link DC, Graubert TA, DiPersio JF, Wilson RK. DNA sequencing of a cytogenetically normal acute myeloid leukaemia genome. Nature. 2008 Nov 6;456(7218):66-72. doi: 10.1038/nature07485. PMID 18987736
- [Background] Miller CA, Wilson RK, Ley TJ. Genomic landscapes and clonality of de novo AML. N Engl J Med. 2013 Oct 10;369(15):1473. doi: 10.1056/NEJMc1308782. No abstract available. PMID 24106950
- [Background] Juliusson G, Antunovic P, Derolf A, Lehmann S, Mollgard L, Stockelberg D, Tidefelt U, Wahlin A, Hoglund M. Age and acute myeloid leukemia: real world data on decision to treat and outcomes from the Swedish Acute Leukemia Registry. Blood. 2009 Apr 30;113(18):4179-87. doi: 10.1182/blood-2008-07-172007. Epub 2008 Nov 13. PMID 19008455
- [Background] Dohner H, Estey E, Grimwade D, Amadori S, Appelbaum FR, Buchner T, Dombret H, Ebert BL, Fenaux P, Larson RA, Levine RL, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz M, Sierra J, Tallman MS, Tien HF, Wei AH, Lowenberg B, Bloomfield CD. Diagnosis and management of AML in adults: 2017 ELN recommendations from an international expert panel. Blood. 2017 Jan 26;129(4):424-447. doi: 10.1182/blood-2016-08-733196. Epub 2016 Nov 28. PMID 27895058